CLINICAL TRIAL: NCT00564993
Title: Cardiac Imaging Under Exercise Stress Test for Early Assessment of Right Ventricular Function in Patients With Tetralogy of Fallot and Pulmonary Regurgitation
Brief Title: Cardiac Function Under Stress for Early Detection of the Right Ventricular Insufficiency After Repair of Tetralogy of Fallot
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MP 4.3 Fallot-stress; EudraCT number: 2007-003461-41
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2011-08

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot | interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): necessary re-intervention (pulmonary valve replacement) after repair of Fallot:
  2 Visits with cardiac imaging under rest and stress (Dobutamin) before and after pulmonary valve replacement
  Interventions: Drug: Dobutamin
- B (Active Comparator): comparison group: with a good result of repair of tetralogy of fallot and good ventricular function:
  1 Visit with cardiac imaging under rest and stress (Dobutamin)
  Interventions: Drug: Dobutamin

INTERVENTIONS:
Drug: Dobutamin — 10&20 µg/kg/min

SUMMARY:
Summary:

The investigators aim to identify markers of right ventricular dysfunction in patients with severe pulmonary regurgitation following repair of Tetralogy of Fallot, that allow prediction of the optimal timing of the replacement of the regurgitant valve. The investigators will use MR as a gold-standard reference for measurement of cardiac function during rest and dobutamine stress. The investigators will also evaluate the predictive potential of tissue Doppler imaging in this patient group.

Purpose:

To predict the optimum timing of pulmonary valve replacement for severe regurgitation in repaired Tetralogy of Fallot using Cardiac Magnetic resonance with dobutamine stress testing.

DETAILED DESCRIPTION:
Tetralogy of Fallot (ToF) is the single commonest complex cardiac condition. It consists of ventricular septal defect (VSD), overriding of the aorta in association with the VSD, pulmonary stenosis and right ventricular (RV) hypertrophy. Surgical repair is indicated as it significantly improves life-expectancy. The results of surgical repair have improved steadily over the last 40 years resulting in a significant population surviving into young adulthood. However, standard repair techniques induce regurgitation of the pulmonary valve due to relief of the right ventricular outflow tract obstruction. Over time this regurgitation induces right ventricular dilatation and dysfunction. RV dilatation and dysfunction correlate with reduced exercise tolerance, arrhythmias, and sudden death following repair.

Replacement of the pulmonary valve, late after primary repair of ToF, has generally been shown to improve symptoms as measured by NYHA classification as it improves haemodynamics, exercise tolerance and dysrhythmia. Though generally safe, surgical replacement of the pulmonary valve exposes the patient to cardio-pulmonary by-pass, which may have detrimental effects on both the myocardium and the brain. Furthermore transplanted valves of various types have a limited life span and thus early repair of the pulmonary valve may instigate a series of re-operations, which will recur throughout the patient's life exposing them to a cumulative risk of morbidity and mortality. Unfortunately there is evidence in the literature that symptomatic improvement is reduced if pulmonary valve replacement is delayed for too long. This is probably due to irreversible myocardial damage with little remodeling of the RV despite a competent pulmonary valve.

In the light of these two opposing factors; potential for failure to recover and avoiding multiple operations there is a need to establish preoperative markers which will allow identification of the failing ventricle before it passes the point of recovery. This will allow close follow-up with intervention timed to minimize loss of function whilst taking into account the likely need for re-operation.

However, it is still unclear, which criteria give the best indication for the need of re-interventions. Two other studies of the Competence Network for Congenital Heart Defects ("Follow up of Post-Repair Tetralogy of Fallot (HP 4.1)" and "Early re-intervention in infants and small children after correction of Tetralogy of Fallot: Prospective analysis of myocardial benefit using cardiac MRI and echocardiography (HP 4.2)" analyze the benefit of such re-interventions and will hopefully provide substantive information on timing of PVR.

There are however references in literature that cardiac imaging procedure under stress possibly results in more sensitive predictive parameters of right ventricular insufficiency than conducted under rest. Dobutamine stress testing has a long history of safe and clinically useful application in ischemic cardiomyopathy and recent studies have demonstrated it's useful predictive value in various outcomes for non-ischemic cardiomyopathy.

Accurate post-operative characterization will allow identification of pre-operative predictive markers. The investigators believe that dobutamine stress testing may in fact be an excellent predictive marker. Dobutamine increases intrinsic contractability as well as reducing after load. It is thought that the failing heart is not able to positively respond to the dobutamine stimulus, and dobutamine stress will thus demonstrate evidence of irreversible damage. Identification of predictive markers of the point at which irreversible myocardial damage occurs will allow better timing of pulmonary valve replacement and will have significant ramifications for the management of this patient group.

In this study imaging procedures (MRI and echocardiography) under rest and stress (dobutamine) are compared before and after pulmonary valve replacement at severe pulmonary insufficiency after repair of Tetralogy of Fallot, whereas the imaging procedure of echocardiography under stress is optional. The data obtained are supposed to determine new parameters of the early right ventricular insufficiency. The investigators will correlate the above objective data with subjective data of change in symptoms and exercise capacity pre- and post-repair. Fallot patients with a good result of repair and good right ventricular function will serve as a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient or patient's legal representatives
* No participation in another AMG driven study within the past 4 weeks or during the whole duration of this study
* Patients with Tetralogy of Fallot after corrective surgery

  * group A (n=45): Adolescents ≥ 14 years or adults with Tetralogy of Fallot after corrective surgery and necessary re-intervention (pulmonary valve replacement because of pulmonary insufficiency
  * group B (n=35): Adolescents ≥ 14 years or adults with Tetralogy of Fallot after corrective surgery and good result of repair and good right ventricular function

Exclusion Criteria:

Non-specific

* pregnancy or lactation
* women of child-bearing age who are sexually active without practising highly effective methods of contraception (a urine/serum pregnancy test may be requested at the discretion of the investigator)
* any diseases or impairment that, in the opinion of the investigator, would justify to exclude a subject from participation
* substance abuse (alcohol, medicines, drugs)
* other medical, psychological or social circumstances that would adversely affect a patient's ability to participate reliably in the study or increase the risk to themselves or others if they participated
* insufficient compliance
* disagreement with storage & transfer of anonymized disease data within this study.
* Persons who are detained officially or legally to an official institution

Specific

* contraindication against pharmacological stress testing (ventricular tachycardia or severe arrhythmia, profound pulmonary stenosis and hypertension of the pulmonary artery)
* coronary heart disease
* atrial fibrillation or flutter
* DORV (if there is another VSD than subaortic)
* associated severe heart defects
* associated other severe (=hemodynamic significantly) valvular defects except for pulmonary insufficiency
* Other clinically relevant diseases, such as malignant tumour or florid diseases (as considered by the investigating physician)
* MRI contraindication, e.g. cardiac pacemaker, implanted neurostimulators and other magnetisable foreign bodies
* Patient is not able to perform spiroergometry (bicycle/treadmill) or existing contraindications
* Patients with Type I or II diabetes
* prohibited concomitant medication: MAO-inhibitors
* Treatment with beta- or alpha-blocker
* Treatment with high doses of ACE-inhibitors or inhibitors of the AT- receptor and permanent treatment with nitrates (in the investigating physician's risk assessment)
* Anticoagulation treatment (risk-benefit decision by the investigating physician, as there may be additional inhibition of platelet aggregation with dobutamine)
* Treatment with diuretics (risk-benefit decision by the investigating physician, as there may be enhancement of the hypokalemia by administration of dobutamine); if necessary verification of the serum K+ -level before exposure to dobutamine
* all contraindications against the study medication described in the SMPC

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Identification of predictive parameters of right ventricular insufficiency | 1 year

SECONDARY OUTCOMES:
Evaluation of mortality, morbidity, pulmonary function, objective exercise tolerance, life-quality and prevalence of cardiac arrhythmia after pulmonary valve replacement | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Beerbaum, MD, Study Chair — Evelina Children's Hospital, Guy's and St. Thomas Foundation Trust, Interdisciplinary Medical Imaging Group, King's College London
Locations (11):
- Germany (11):
  - Universitätsklinikum Freiburg, Klinik III Päd. Kardiologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Klinik für Kinderheilkunde und Jugendmedizin, Tübingen, Baden-Wurttemberg
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Medizinische Hochschule Hannover, Pädiatrische Kardiologie und Intensivmedizin, Hanover, Lower Saxony
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Klinik und Poliklinik für Kinder- und Jugendmedizin, Pädiatrische Kardiologie, Münster, North Rhine-Westphalia
  - Deutsches Kinderherzzentrum St. Augustin, Sankt Augustin, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg/Saar, Saarland
  - Herzzentrum Leipzig, Klinik für Kinderkardiologie, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Deutsches Herzzentrum Berlin, Berlin, State of Berlin

REFERENCES:
- See also: Competence Network for Congenital Heart Defects — http://www.kompetenznetz-ahf.de